CLINICAL TRIAL: NCT04896970
Title: Risk of SARS-CoV-2 Infection in a Standing Concert in a Closed Performance Hall
Brief Title: Risk of SARS-CoV-2 Infection (COVID-19) in a Standing Concert in a Closed Performance Hall
Acronym: ConcerTest
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: abandonment
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RECHMPL21_0110
Record Dates: First submitted 2021-05-11; First posted 2021-05-21 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: SARS-CoV-2
Keywords: SARS-CoV-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concert (Experimental): Participants will go to a concert in a closed hall.
  Interventions: Other: Concert
- Control (No Intervention): Participant will stay at home.

INTERVENTIONS:
Other: Concert — A musical show in a closed hall, lasting for about 2 hours, in respects of safety measure (masks, hydroalcoholic gel, etc…) with approximately 200 participants.
  Arms: Concert

SUMMARY:
The investigators want to compare the SARS-CoV-2 incidence 7 days after having been screened negative, between two groups of adults randomized to either go to a concert or not.

Participants will be screened via a rapid saliva test a few hours before the show. The hypothesis is that attending a standing concert in respect of safety precaution doesn't increase the risk of SARS-CoV-2 infection.

DETAILED DESCRIPTION:
Context :

A previous Spanish randomized study in November 2020 concluded in a non superiority of the SARS-CoV-2 incidence in RT-PCR-negative participant of a concert compared to a control group. In the same way, investigators want to compare the SARS-CoV-2 incidence of participants of a concert 7 days after the show with a control group, using a saliva test.

While naso-pharyngeal RT-CPR is the gold-standard for virological SARS-COV-2 tests, this method can be painful and results take time. Saliva rapid tests have satisfactory diagnostic performances and easy access to results. Saliva rapid tests may lead to mass screening in cultural mass events.

This project has the specific feature to be set in closed concert hall with limited size attendance.

Methodology :

This experimental monocentric randomized non-inferiority will compare 2 parallel groups (with single blind for the screening tests results). The randomization will be centralised and stratified on the age.

Program :

Participants will be informed via an information notice and a preselection screening questionnaire on the internet. Eligible participants will have to come on the day of the show near the concert place to be included (after information and signing of the consent form). participants will receive a saliva sample tube.

Positively screened participants will have to go home. The others will be randomized in two groups. Participants will both have to come back 7 days after for the second screening.

Feasibility :

The concert place have a strong fan base to recruit participants from. To include all the participants, two concerts will take place, separated by a few days. Participants will receive goodies to maximize the chance of them attending to both screening.

This project received a methodological support from the Clinical and Epidemiological Research Unit of the Montpellier Hospital and is promoted by the Montpellier Hospital.

Sys2diag and SkillCell which developed the screening tests are involved as well as VOGO for the technical part and data management.

This project is financially helped by Région Occitanie, Montpellier Métropole, Saint-Jean-de-Vedas, SACEM, APEM, Tout à Fond and Boomerang.

ELIGIBILITY:
Inclusion criteria:

* At least 18 and less than 60 years old
* Having completed the internet pre selection questionnaire and signed the consent form
* Negative rapid saliva RT-LAMP EasyCov test on the day of the show
* Social Security Affiliation

Exclusion criteria:

* Serious form Covid-19 risk factors
* Positive saliva rapid test on the day of the event (and people who came with a positive person)
* History of SARS-CoV-2
* SARS-CoV-2 vaccination
* Living with a person older than 75 years old or having a serious form of Covid-19 risk factor
* Protection of a legal conservator
* Pregnant or breastfeeding women
* People living with a pregnant or breastfeeding woman

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV-2 incidence | 7 days after the first screening
  Rate of newly SARS-CoV-2 infected participants

SECONDARY OUTCOMES:
Time to screen all participants | At screening day
  time spent to screen and have results for every participant of the concert